CLINICAL TRIAL: NCT02215538
Title: Concerta in the Treatment of Adult ADHD and a Comparison of Four Adult ADHD Scales and Effects on Personality
Brief Title: OROS Methylphenidate (Concerta) in the Treatment of Adult ADHD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, frederick reimherr, Director, Mood Disorders Clinic, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 00012246
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; adult; WRAADDS; OROS MPH; emotional dysregulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OROS methylphenidate (Experimental): This was a 4-week double-blind arm. Medication was initiated at 18 mg/day and increased every 2 or 3 days by 9 mg based on treatment response and side effects. Maximum dose - 90 mg/day. Patients were seen weekly. Generally a stable dose was seen in 2 weeks and maintained the last 2 weeks of the arm. Side effects were assessed at each visit.
  Interventions: Drug: OROS methylphenidate
- placebo (Placebo Comparator): This arm was identical to the active medication arm except that placebo replaced the active medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OROS methylphenidate
  Other Names: concerta
  Arms: OROS methylphenidate
Drug: Placebo — Placebo medication appears identical to the active medication OROS methylphenidate
  Arms: placebo

SUMMARY:
This study will look at the effectiveness of osmotic release oral system (OROS) methylphenidate (Concerta) in treating attention deficit hyperactvity disorder (ADHD) in adults. Concerta has received FDA approval for childhood ADHD and there is documentation that it is effective in adult ADHD. However this trial will explore its effectiveness in treating symptoms not a part of the Diagnostic and Statistical Manual-III (DSM-III) criteria. Subjects will experience one screening visit and one baseline visit. Those who meet admission criteria will enter the double-blind phase. This will involve two 4-week treatment periods one of which will involve the use of Concerta and the other a placebo pill. Subjects who complete the double-blind phase will be allowed to enter a 180-day, open-label Concerta phase designed to assess long-term effects.

DETAILED DESCRIPTION:
ADHD affects from 3 to 5% of children, persists into adolescence 40 to 70% of these children and continues into adulthood in at least 50% of affected adolescents. Pharmacotherapy for ADHD in adults has paralleled that used for children, with generally positive results (Spencer, 1998). Never-the-less, it is not clear that the dimensions of medication response in adults are the same as in children. The extent to which the symptoms change with age remains open to question. This trial is created to include a variety of outcome measures which will enhance the number of symptoms assessed.

Methylphenidate was the first medication shown to be effective in treatment for adults with ADHD and continues to be widely used. Several studies have demonstrated the usefulness of methylphenidate in adult ADHD (Wender et al, 1985, Spencer et al, 1995). These studies have not shown any unexpected drawbacks to treatment with methylphenidate. The extended release formulations represent an improvement over the immediate release versions for many patients.

This is a double-blind, placebo-controlled, randomized, crossover trial comparing OROS methylphenidate with placebo. The double-blind trial will be preceded by an enrollment period consisting of a screening visit followed by a baseline visit. Patients who continue to meet admission criteria at baseline will be randomized into the first of two 4-week treatment periods. We will attempt to reach the highest tolerated dose size within 2 weeks and then observe the response over the last two weeks of each crossover phase. The double-blind period will be followed by a 180 day open-treatment, flexible-dose phase designed to assess long-term effects.

ELIGIBILITY:
Inclusion Criteria:

Adults meeting DSM-IV-Text Revision criteria for ADHD, the Utah Criteria for ADHD, and experiencing at least moderate impairment (a score of 4 or greater on the CGI-Severity Scale for ADHD at both Screening and Baseline visits) will be enrolled. Other criteria include:

1. Subjects ages 18 to 65, inclusive;
2. Female subjects are eligible to enter and participate in this study only if:

   * She is of non-childbearing potential; has a male sexual partner who is surgically sterilized; is on implant of levonorgestrel, injectable progesterone, or an oral contraceptive; has an intrauterine device (IUD); or is sexually inactive with a male partner.
   * Or agrees to use a double barrier method of contraception (any combination of physical and chemical methods) and has a negative urine pregnancy test at screening interview.
3. Subject must be in general good health as determined by medical history, ECG, and other analysis that, in the judgment of the study physician, would confirm the patient's good health.
4. Subjects must read and write at a level sufficient to provide written informed consent and complete study-related materials.

Exclusion Criteria:

1. Subjects with other current DSM-IV Axis I Disorders including Current or lifetime history of psychosis, current bipolar disorder type I, current Major Depressive Disorder, and Current Anxiety Disorder (unless in the opinion of clinic physician ADHD is the primary disorder and causes the disability seen in the patient);
2. Subjects with any other DSM-IV Axis II diagnosis so severe that it would suggest non-responsiveness to pharmacotherapy for ADHD or noncompliance with the protocol;
3. Subjects at risk for suicide or a risk to harm others;
4. History of Substance Dependence according to DSM-IV criteria within 3 months of screening;
5. Subjects currently abusing illegal drugs or alcohol are excluded from the study;
6. Positive urine screen for drugs of abuse at screening for patients who have a significant history of substance use but still meet criteria 4 and 5. Patients not at risk for substance abuse will not be given a urine drug screen;
7. Subjects in whom stimulants would represent a risk such as those with a history of stimulant abuse,
8. History of uncontrolled hypertension or significant cardiovascular disease;
9. Any known or suspected significant medical or psychiatric illnesses (e.g., hepatic or renal insufficiency, pulmonary (asthma, chronic obstructive pulmonary disease, etc), gastrointestinal, endocrine, neurological or metabolic disturbances that, in the judgment of the investigator, may impair interpretation of study results or constitute a significant safety concern in the context of the clinical trial;
10. Medications, including health food supplements judged by the investigator to be likely to have central nervous system activity (for example, St John's Wort, gingko leaf, and melatonin), are not permitted during the study. If the subject is taking the medication prior to study entry, there must be a 7 day washout period prior to Visit 2. We will ask for an honest report of all medications consumed between visits. In the event a medication with psychoactive properties is consumed, the patient will be counseled regarding the use of prohibited medications;
11. Use of any medication not considered acceptable by the clinical investigator or the medical monitor during the 7-day period before the start of the study (Day 1);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-11; Primary Completion 2006-02 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Wender-Reimherr Adult Attention Deficit Disorder Scale (WRAADDS) | Baseline visit, Double-blind phase Week 4 each arm, Open-Label months 1-6
  This is an investigator rated scale which assessed the 7 domains of the Utah Criteria of Adult ADHD

SECONDARY OUTCOMES:
Clinical Global Impressions-Improvement (CGI-I) | Baseline; Double-blind phase Week 4 each arm: Open-Label months 1-6
  This is a global measure in improvement in symptoms that is a Likert type scale
Clinical Global Impression - Severity (CGI-S) | Baseline visit; Double-blind phase Week 4 each arm: Open-Label months 1-6
  This is a general measure of symptom severity assessed using a Likert type scale.
ADHD rating scale (ADHD-RS) | Baselinevisit; Double-blind phase Week 4 each arm: Open-Label final visit month 6
  This is an investigator rated scale which assesses the DSM-IV symptoms.
Self Report Wender-Reimherr Adult Attention Deficit Disorder Scale (SR-WRAADDS) | Baseline; Double-blind phases Week 4 each arm: Final visit of Open-Label period month 6
  This is a patient rated scale that assesses the 7 domains of the Utah Criteria for adult ADHD as well as ODD, Social functioning and Learning difficulties.
Wisconsin Personality Inventory - IV (WISPI-IV) | Baseline visit; Final Open-Label visit month 6
  This is a computerized personality inventory completed by the patients. It consists of 214 items which address the 10 DSM-IV personality disorders plus passive aggressive personality disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick W Reimherr, MD, Principal Investigator — Univeristy of Utah Dept of Psychiatry
Locations (1):
- Mood Disorders Clinic, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Marchant BK, Reimherr FW, Halls C, Williams ED, Strong RE. OROS methylphenidate in the treatment of adults with ADHD: a 6-month, open-label, follow-up study. Ann Clin Psychiatry. 2010 Aug;22(3):196-204. PMID 20680193
- [Result] Reimherr FW, Marchant BK, Williams ED, Strong RE, Halls C, Soni P. Personality disorders in ADHD Part 3: Personality disorder, social adjustment, and their relation to dimensions of adult ADHD. Ann Clin Psychiatry. 2010 May;22(2):103-12. PMID 20445837
- [Result] Robison RJ, Reimherr FW, Gale PD, Marchant BK, Williams ED, Soni P, Halls C, Strong RE. Personality disorders in ADHD Part 2: The effect of symptoms of personality disorder on response to treatment with OROS methylphenidate in adults with ADHD. Ann Clin Psychiatry. 2010 May;22(2):94-102. PMID 20445836
- [Result] Williams ED, Reimherr FW, Marchant BK, Strong RE, Halls C, Soni P, Gale PD, Robison RJ. Personality disorder in ADHD Part 1: Assessment of personality disorder in adult ADHD using data from a clinical trial of OROS methylphenidate. Ann Clin Psychiatry. 2010 May;22(2):84-93. PMID 20445835
- [Result] Reimherr FW, Williams ED, Strong RE, Mestas R, Soni P, Marchant BK. A double-blind, placebo-controlled, crossover study of osmotic release oral system methylphenidate in adults with ADHD with assessment of oppositional and emotional dimensions of the disorder. J Clin Psychiatry. 2007 Jan;68(1):93-101. doi: 10.4088/jcp.v68n0113. PMID 17284136
- [Derived] Gift TE, Reimherr FW, Marchant BK, Steans TA, Wender PH. Personality Disorder in Adult Attention-Deficit/Hyperactivity Disorder: Attrition and Change During Long-term Treatment. J Nerv Ment Dis. 2016 May;204(5):355-63. doi: 10.1097/NMD.0000000000000470. PMID 27082828